CLINICAL TRIAL: NCT01439828
Title: Randomized and Double-blind Clinical Trial of N-acetylcysteine Versus Placebo Efficacy in the Cannabis Withdrawal
Brief Title: Clinical Trial of N-acetylcysteine Versus Placebo Efficacy in the Cannabis Withdrawal
Acronym: MUCOCRAV
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P081120
Record Dates: First submitted 2011-09-21; First posted 2011-09-23 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2012-01

CONDITIONS: Cannabis Dependence; Cannabis Abuse
Keywords: Cannabis; N-Acetylcystein; Dependence; Abuse; Craving; Genetic
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental : N-acetylcystein (Experimental): N-acetylcystein and placebo doses will be increased if craving decreases <25% compared to the previous visit. The doses start at 200 mg x 4/24h to 800 mg x 4/24h
  Interventions: Drug: N-acetylcystein
- Placebo Comparator (Placebo Comparator): N-acetylcystein and placebo doses will be increased if craving decreases <25% compared to the previous visit. The doses start at 200 mg x 4/24h to 800 mg x 4/24h
  Interventions: Drug: N-acetylcystein

INTERVENTIONS:
Drug: N-acetylcystein — Visit 1: Consent signed. Blood and urine analysis. Questionnaires assessing cannabis and tobacco's craving.N-acetylcystein and placebo doses will be increased if craving decreases <25% compared to previous visit.The doses start at 200 mg x 4/24h to 800 mg x 4/24h.Visit 2 to 5: Medication safety and cannabis craving and withdrawal assessment during 4 weeks.

SUMMARY:
The primary purpose is to assess the efficacy in human of N-acetylcysteine versus placebo during 4 weeks in cannabis withdrawal.

DETAILED DESCRIPTION:
Introduction:There are few clinical trials on pharmacotherapies in marijuana dependence. There is no randomized and double-blind trial on N-acetylcysteine efficacy in marijuana withdrawal.Aims:The first aim is to assess the efficacy in human (n=150 outpatients) of N-acetylcysteine versus placebo during 4 weeks in cannabis withdrawal.The secondary aims are:a-Assessing the abstinence during the next 5 months of follow-up.b-Assessing the correlations between genetic characteristics: cytochrome CYP2C9 and CYP3A4, CNR1 receptor, Fatty Amide Hydroxylase (FAAH), dopamine DAT transporters and Catechol-O-MéthylTransférase (COMT); and three phenotypes : 1. cannabis level consumption, 2. cannabis abuse and dependence (DSM-IV), and 3. cannabis withdrawal.c-Assessing tobacco consumption (Fagerström test), NICOTINIQUE receptor CHRA3 and cannabis quitting success.Subjects:150 cannabis outpatients, seeking treatment in LARIBOISIERE hospital cannabis setting, to cut down their cannabis use.Inclusion criteria: > 18 year old, not pregnant or breast feeding, cannabis abuse or dependence diagnosis (DSM-IV), acceptance of the trial and consent signed, validated by ethic committee.Methods:Randomized and double-blind trial.Visit 0: Clinical assessment and trial presentation, Validate inclusion and non- inclusion criteria.Visit 1: Consent signed. Blood and urine analysis. Questionnaires assessing cannabis and tobacco's craving.NAC and placebo doses will be increased if craving decreases <25% compared to previous visit. The doses start at 200 mg x 4/24h to 800 mg x 4/24h.Visit 2 to 5: Medication safety and cannabis craving and withdrawal assessment during 4 weeks.Visit 5: Blood and urine analysis.Visit 6 to 8: abstinence assessment during 5 months.Goals:Efficacy assessment of N-Acetylcysteine in cannabis withdrawal and abstinence compared to placebo. Assessment of NAC efficacy in cannabis craving. The length of the study is 6 months to evaluate abstinence persistence. Evaluation of clinical, biological and genetic factors associated with abstinence success.Statistic :Sample size : A two group continuity corrected c2 test with a 0.050 two-sided significance level will have 80% power to detect the difference between a Group 1 proportion, p1, of 0.250 and a Group 2 proportion, p2, of 0.500 (odds ratio of 3.000) when the sample size in each group is 66. Taking into account a rate of lost of follow-up around 15 % the total sample size of the study has been fixed at N= 150 patients.Main criterion and binary secondary criteria will be analysed by Chi-square tests or Fisher's exact probability test. Relationships between genotype and phenotypes will be analysed by multivariate logistic models

ELIGIBILITY:
Inclusion Criteria:

* > 18 year old
* Not pregnant or breast feeding
* Cannabis abuse or dependence diagnosis (DSM-IV)
* Acceptance of the trial and consent signed, validated by ethic committee
* Patient affiliated to social insurance care

Exclusion Criteria:

* Contraindication to N-acetylcystein : allergic to N-acetylcystein, severe allergic illness, PHENYLCETONURIA, lactose intolerance, gastro-duodenal ulcer.
* Severe somatic disease not stabilized : diabetes, epilepsia, recent myocardial infarcts, asthma.
* Severe mental disease not stabilized : schizophrenia.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2012-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Success rate of withdrawal defined by a reduction of at least 50% of the rate of urinary carboxy-THC | at 4 weeks

SECONDARY OUTCOMES:
The success rate of withdrawal defined by a declarative reduction of at least 50% of the cannabis | at 2, 3 and 6 months
The retention rate of withdrawal | at 6 months
The rate of complete cessation of cannabis use | at 4 weeks and 2, 3 and 6 months.
  Declarative clinical criteria by the patient and validated at D28 by the decrease of at least 50% of the report of the dosage of the report CarboxyTHC / creatinine
Phenotypic profile (3 major types) | at Day 28 (end of treatment)
  * The amount of cannabis and THC consumed with use of the upper quartile to define a high consumption and the lowest quartile to define the weak consumer
  * Dependence and abuse according to DSM IV criteria;
  * Withdrawal syndrome in dependent patients according to DSM IV and the scale of MJQQ Gorelick.

CONTACTS AND LOCATIONS:
Overall Officials: Eric GUILLEM, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Psychiatrie - Hôpital Lariboisière, Paris, France